CLINICAL TRIAL: NCT04318821
Title: Effect of Laser Acupuncture on Adhesive Small Bowel Obstruction: a Prospective Double-blind Randomized Controlled Trial
Brief Title: Effect of Laser Acupuncture on Adhesive Small Bowel Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8K0571
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-07

CONDITIONS: Adhesive Small Bowel Obstruction
Keywords: Adhesive small bowel obstruction; Laser acupuncture; Acupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The participants in each group will receive real (with energy output) or sham (without energy output) laser acupuncture. The feelings of participants in each group are not different. The care provider and outcomes assessor don't involve the random allocation and don't know if participants receive real laser acupuncture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LA group (Experimental): The subjects in the experimental group will receive 0.375 J of energy at each of the following acupoints: LI4 (Hegu, B3), PC6 (Neiguan, B3), ST25 (Tianshu, B3), ST36 (Zusanli, B2), CV4 (Guanyuan), CV12 (Zhongwan, B3).
  Interventions: Procedure: Laser acupuncture
- Control group (Sham Comparator): The subjects in the control group will receive sham LA treatment, without any laser output (no stimulation) at the same acupoints used in experimental group.
  Interventions: Procedure: Laser acupuncture

INTERVENTIONS:
Procedure: Laser acupuncture — Laser acupuncture is a non-invasive therapy that involves stimulation of traditional acupoints with low-intensity, non-thermal laser irradiation.

SUMMARY:
Adhesive small bowel obstruction (ASBO) is one of the most common complications and is a major cause of admission after intra-abdominal surgery. To date, the ideal management of ASBO remains controversial. The aim of this protocol designed as a double-blind randomized controlled trial is to investigate the efficacy of laser acupuncture (LA) therapy in patients with ASBO.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 80 years
* Clinical symptoms and signs of mechanical obstruction

Exclusion Criteria:

* Clear non-adhesive etiology of small bowel obstruction (e.g. tumor, hernia)
* Emergency surgical intervention before being admitted to the hospital
* Pregnancy
* Local skin infection on the acupoints, and limb amputees.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Success rate of conservative treatment | 2 week
  Defined as no need for long term nasogastric tube decompression and operative intervention.

SECONDARY OUTCOMES:
Time to oral intake | 2 weeks
  Defined as participants can try intake due to symptoms improved including nausea, vomiting, distension and pain.
Length of hospital stay | Through study completion, an average of 1 year
  Date from admission to discharge
Serum lipase | Up to 2 weeks
  Serum lipase
Serum amylase | Up to 2 weeks
  Serum amylase
Serum cortisol | Up to 2 weeks
  Serum cortisol
Serum motilin | Up to 2 weeks
  Serum motilin
Serum ghrelin | Up to 2 weeks
  Serum ghrelin
Serum intestinal fatty acid binding protein (I-FABP) | Up to 2 weeks
  Serum intestinal fatty acid binding protein (I-FABP)

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ting Liu, MD, Principal Investigator — Department of Chinese Medicine, Kaohsiung Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shih CH, Hsieh TM, Wu BY, Liu CT. Effect of laser acupuncture on adhesive small bowel obstruction: A prospective double-blind randomized controlled trial. Medicine (Baltimore). 2021 Mar 5;100(9):e25035. doi: 10.1097/MD.0000000000025035. PMID 33655978